CLINICAL TRIAL: NCT02127645
Title: PILOT OBSERVATIONAL STUDY OF NEOADJUVANT 5 x 5 RADIOTHERAPY FOLLOWED BY TRANSANAL ENDOSCOPIC MICROSURGERY FOR T1-T2 EXTRAPERITONEAL RECTAL CANCER WITH CURATIVE INTENT
Brief Title: Neoadjuvant Radiotherapy Followed by Transanal Endoscopic Microsurgery for T1-T2 Extraperitoneal Rectal Cancer
Acronym: NERATEM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Association for Endoscopic Surgery (Other)
Responsible Party: Principal Investigator, Alberto Arezzo, Assistant Professor of Surgery, European Association for Endoscopic Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EAES-4
Record Dates: First submitted 2014-04-26; First posted 2014-05-01 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: RECTAL CANCER
Keywords: RADIOTHERAPY; TRANSANAL ENDOSCOPIC MICROSURGERY; LOCAL EXCISION
MeSH Terms: conditions — Rectal Neoplasms | interventions — Transanal Endoscopic Microsurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Early Rectal Cancer (Experimental): patients with T1 - T2, N0, G1-2 rectal cancer
  Interventions: Procedure: SRT-TEM; Procedure: LRT-TEM; Procedure: Transanal Endoscopic Microsurgery (TEM); Procedure: Total Mesorectal Excision (TME)

INTERVENTIONS:
Procedure: SRT-TEM — SRT-TEM underwent 25 Gy RT followed by TEM
  Other Names: Transanal Endoscopic Microsurgery (TEM); Neoadjuvant Short course Radio-Therapy
Procedure: LRT-TEM — TEM following 46 Gy RT
  Other Names: Transanal Endoscopic Microsurgery (TEM); Neoadjuvant Long Term Radio-therapy 46 Gy
Procedure: Transanal Endoscopic Microsurgery (TEM) — Transanal Endoscopic Microsurgery (TEM)
Procedure: Total Mesorectal Excision (TME) — Laparoscopic Total Mesorectal Excision
  Other Names: Laparoscopic Total Mesorectal Excision

SUMMARY:
Objective: Recent randomized and non-randomized studies suggest that neoadjuvant radiotherapy followed by Transanal Endoscopic Microsurgery (TEM) show comparative results to abdominal resection in pT2 extraperitoneal cancer. As the risk of lymphnode metastases is significant already for T1 invasive cancers with submucosa infiltration >1 mm it is our intention to investigate in both T1sm2-3 and T2 rectal adenocarcinomas the effectiveness of this combined treatment in a case series comparing results of this pilot study to an historical series of patients affected by T1-T2 rectal cancer who underwent anterior resection (AR) or total mesorectal excision (TME) with or without abdomino-perineal resection (APR) with no neoadjuvant therapy.

If equally effective, TEM offers a further reduction in invasiveness of treatment, which should correspond to a lower morbidity, mortality and a better quality of life.

DETAILED DESCRIPTION:
Study design: This is a single centre case series pilot study which oncologic results will be compared to historical data collected consisting of patients treated by anterior resection (AR) or total mesorectal excision (TME) with or without abdomino-perineal resection (APR) with no neoadjuvant radiotherapy.

Study population: Patients with T1sm2-3 and T2, N0, G1-G2, located between 2 and 12 cm from the anal verge, in a health condition that permits general anesthesia.

Interventions: Neoadjuvant radiotherapy at a dose of 25 Gy (5 Gy per day for 5 consecutive days) is administered to the patient. Within 10 days after the end of radiotherapy TEM will be performed.

Primary Endpoint: incidence of recurrence at 36 months

Primary outcome measure (for non-inferiority):

Local recurrence of neoplasia, defined as the presence of histologically proven neoplastic tissue in either visible recurrent lesions or in random biopsies, taken at surveillance endoscopies after the intervention strategy has been completed. Patients will undergo surveillance endoscopies at 3, 6, 12, 18, 24 and 36 months by an independent endoscopist. During each surveillance endoscopy local recurrence will objectively be defined by the Higaki criteria for recurrence: tumor appearing within a clear resection scar; tumors with convergent folds; and tumors nearby a clear resection scar (within 5 mm) (39). Targeted biopsies will be taken for histological confirmation; in case of an apparently healed normal scar without evidence of recurrence, biopsies will be taken from the basis and 3 from the edges of the scar to detect occult recurrent neoplasia.

Loco-regional recurrence will be investigated by MRI (CT when MRI contraindicated) which will be performed at 6, 12, 24 and 36 months. Distant metastases will be investigated by standard follow-up according to local policy.

Additional outcome measures:

1. Complications: subdivided into procedural (during treatment) and delayed complications (after ending the procedure); and further subdivided into major (requiring additional surgery) and minor (requiring endoscopic or medical intervention) complications.

   During admission patients will be monitored for complications. The following standardized discharge criteria will be applied: normal intake of nutrition; normal mobility; absence of fever (<38°C); and stable hemoglobin level during 1 day (<1 mmol/L) in case of rectal blood loss. Two weeks after the intervention, a research fellow will contact the patient by telephone again and ask for occurred complications.
2. Generic and disease-specific health related quality of life will be measured at baseline, 2 weeks, 3 months, 6 months, 1 and year follow-up by the SF-36, EORTC Q30, EORTC Q38 and Wexner score (for incontinence) questionnaires.
3. Measurement of anorectal functional outcome by anal manometry and rectal volumetry (barostat) before and 3 months after treatment.

Sample size: As a pilot study, sample size is not available

Economic evaluation: A cost-effectiveness and cost-utility analysis of neoadjuvant RT followed by TEM for extraperitoneal rectal cancer with respectively the costs per recurrence free patient and the cost per quality adjusted life year as primary outcome measures, compared to the historical series of patients who underwent surgery without neoadjuvant radiotherapy, will be performed.

Time schedule: 36 months for inclusion (June 1st 2011 - May 31st 2014), 36 months minimum follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a large rectal sessile or flat lesion (type 0-Is, 0-II or 0-III according to the Paris Classification) with the largest diameter of 2 cm or larger11 (estimated by an opened resection snare).
* lower and upper borders of the rectal neoplasm located between 2 and 12 cm from the anal verge, respectively.
* Biopsies of the lesion showed neoplastic tissue adenocarcinoma G1-G2 on histopathological evaluation.
* Endoscopic ultrasonography (EUS) of the rectal lesion confirmed invasion into the submucosal layer (uT1sm) >1 mm or the muscle layer (uT2) and ruled out the presence of lymph nodes >1 cm.
* Pelvic Magnetic Resonance Imaging (MRI) (or Computer Tomography (CT) when MRI was contraindicated) ruled outlymph nodes >1 cm.
* ASA (America Society of Anesthesiologists)- status I-III.

Exclusion Criteria:

* previous anorectal surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
incidence of local and distant recurrence | 36 months

SECONDARY OUTCOMES:
morbidity, subdivided into major (requiring surgery) and minor (requiring endoscopic or medical intervention) | 30 days
disease specific and general quality of life | 30 days
anorectal function | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Arezzo, Assistant Professor of Surgery, Principal Investigator — European Association of Endoscopic Surgery
Locations (1):
- Department of Surgical Sciences, University of Torino, Turin, Piedmont, Italy